CLINICAL TRIAL: NCT05402306
Title: The Feasibility and Efficacy of a Two-week MCT Treatment of Anxiety Disorders in a Group Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Sverre Urnes Johnson, Associate Professor Sverre Urnes Johnson, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK269896
Record Dates: First submitted 2022-02-28; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Anxiety Disorders
Keywords: Metacognitive therapy; Attention training technique
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): A two-week intensive group treatment with MCT mainly focusing on attention training. The participants will be allocated into treatment in groups of six. Group sessions will be conducted two times a day for approximately 60 minutes.
  Interventions: Other: Treatment group
- Waitlist control group (No Intervention): Cohorts of 12 included patients will be randomly assigned to active treatment or waitlist for two weeks. The waitlist patients will receive the same treatment immediately after four-week waiting period.

INTERVENTIONS:
Other: Treatment group — Group metacognitive therapy, mainly with attention training technique over two weeks.
  Arms: Treatment group

SUMMARY:
Long treatment durations may not always be feasible for patients due to pressure to get better quickly, long travel distance to treatment clinics, inflexible working hours, or childcare. To overcome these challenges intensive treatments are currently emerging and several research studies have shown significant and lasting results of diagnosis-specific intensive treatments. A transdiagnostic treatment in a group setting can contribute to a more efficient course of treatment for patients.

Research suggests that Metacognitive Therapy (MCT) is an effective treatment for anxiety disorders. However, MCT has not previously been used on inpatients over a two-week period. To make the treatment tangible for patients and easy to administer for therapists over a short time, attention training technique (ATT) will mainly be used as a changing technique.

The main aim of the study is to explore the feasibility and efficacy of intensive and short-term MCT for anxiety disorders in a group setting.

DETAILED DESCRIPTION:
Design: The study will use randomized control trial with a waitlist control. Cohorts of 12 included patients will be randomly assigned to active treatment or waitlist for two weeks. The waitlist patients will receive the same treatment immediately after the two-week waiting period.

Inclusion criteria: Adults ranging from 18 to 30 years of age meeting diagnostic criteria for generalised anxiety disorder, social phobia, and/or panic disorder with or without agoraphobia will be included in the study. Further the participants must be able to communicate in Norwegian and provide written consent.

Exclusion criteria: Exclusion criteria will be ongoing drug abuse, history of psychotic episodes, current suicidality, or participants not able to adapt to an intensive group format.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 30 years
* Meeting diagnostic criteria for generalised anxiety disorder, social phobia, and/or panic disorder with or without agoraphobia
* Provide written consent to partake in the study

Exclusion Criteria:

* Ongoing drug abuse
* History of psychotic episodes
* Current suicidality
* Participants not able to adapt to an intensive group format

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-01-28 (Estimated); Study Completion 2023-01-28 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  The Generalized Anxiety Disorder-7 (GAD-7, Spitzer et al., 2006) will be used to measure anxiety symptoms. GAD-7 is a seven-item, self-report measure which assess the severity of anxiety symptoms within the last two weeks. The items are scored on a four-point Likert scale (0-3), with the scores ranging from minimum 0 to maximum 21. Higher scores means worse outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) will be used to measure symptoms of depression. The questionnaire consists of nine items where each is scored on a four-point Likert scale (0-3), with the range of scores from 0 to 27. Higher scores indicate greater depression severity
Social Phobia Inventory (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  Social Phobia Inventory (SPIN; Connor et al., 2000) will be used to measure symptoms of social phobia. SPIN is a 17-item, self-report measure which assess social phobia symptoms during the last weeks. Items is rated from 0 to 4, from "not at all", "a little bit", "somewhat", "very much" to "extremely". The score ranges from 0 to 68. Higher scores indicate greater social anxiety severity. A cut-off score of 19 assumes to indicate a clinical social phobia.
CAS-1 (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  CAS-1 (Wells, 2009) is a 16-item self-report measure which assess metacognitive strategies and metacognitive beliefs within the last week.The first two items examine time used on worry/rumination and threat monitoring rated on an eight-point scale from "no time" to "all the time". The next six items assess unhelpful coping behaviours on the same likert-scale. The last eight items investigate metacognitive beliefs which is rated from 0 to 100. Higher scores means more time spent on CAS and higher belief in metacognitions.
Inventory of Interpersonal Problems (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  Inventory of Interpersonal Problems (IIP-32; Horowitz et al., 2000) is a 32-item self-report questionnaire which measure interpersonal functioning in total and on eight different subscales. The items are rated from 0 "not at all" to 4 "extremely". High scores for the total score and the subscales indicate an increased level of interpersonal problems.
Metacognition questionnaire 30 (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  The Metacognition questionnaire (MCQ-30; Wells & Cartwright-Hatton, 2004) will be used to measure metacognitive beliefs. MCQ-30 is a 30-item self-report measuring general belief in different metacognitions on a scale from 1 to 4, and the responses are "do not agree", "agree slightly", "agree moderately", and "agree very much". The items are divided in five subscales; cognitive confidence, positive beliefs about worry, cognitive self-consciousness, negative beliefs about uncontrollability and danger, and need to control thoughts. The scores for each subscale range from 6 to 24. Summing each subscale gives an overall total score that ranges from 30 to 120, with higher scores indicating higher beliefs in metacognitions.
The Short Warwick-Edinburgh Mental Well-Being scale (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS; Stewart-Brown et al., 2009) is a measure of mental well-being. SWEMWBS is a seven-item self-report related to positive aspects of subjective well-being and psychological functioning over the previous two weeks. Items is rated from 1 "none of the time" to 5 "all of the time". Scores range from 7 to 35 and a higher score indicates a higher level of mental well-being.
Work ability score (WAS) (Change) | Change from baseline; pre-intervention; after the intervention; 3 months follow up; 6 months follow up.
  The single-item Work Ability Score (WAS) will be used to measure work ability. The WAS concerns the first item of the 7-item Work Ability Index (WAI), "Current work ability compared with the lifetime best" (Ilmarines, 2007). The item is rated from 0 "completely unable to work" to 10 "work ability at its best". Higher score indicate greater work ability.

OTHER OUTCOMES:
Ecological Momentary Assessment-questions | 4 times per day before, during and after treatment. The collection will go on for a total of six weeks.
  Single item questions capturing anxiety and depression symptoms, and different mechanisms of change.
Mini-International Neuropsychiatric Interview | Evaluation at baseline, two weeks after the intervention and follow up at 6 months.
  Mini-International Neuropsychiatric Interview (M.I.N.I.; Sheehan et al., 1998) will be used for diagnostic evaluation of the participants.
ADIS Severity Scale in Anxiety Disorders Interview Schedule IV (Brown, DiNardo & Barlow, 1996) | Evaluation at baseline, two weeks after the intervention and follow up at 6 months.
  We will use the ADIS Diagnostic severity Scale to evaluate the severity of the diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo & Modum Bad; Henrik Nordahl, PhD, Principal Investigator — Norwegian University of Science and Technology; KariAnne Vrabel, PhD, Principal Investigator — Modum bad & University of Oslo; Asle Hoffart, PhD, Principal Investigator — Modum Bad & University of Oslo; Therese R. Snuggerud, Masters, Principal Investigator — Modum Bad
Locations (1):
- Modum Bad, Vikersund, Norway

IPD SHARING:
Plan to Share IPD: No